CLINICAL TRIAL: NCT00326820
Title: Zoledronate Versus Ibandronate Comparative Evaluation: A Randomized Phase III, Open-Label, Multicenter, Parallel Group Clinical Trial to Evaluate and Compare the Efficacy, Safety Profile and Tolerability of Oral Ibandronate Versus Intravenous Zoledronate in the Treatment of Breast Cancer Patients With Bone Metastases
Brief Title: Ibandronate or Zoledronate in Treating Patients With Newly Diagnosed Bone Metastases From Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wales Cancer Trials Unit (Other)
Collaborators: Velindre NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000478864; WCTU-ZICE; NCRI-ZICE; ROCHE-ZICE; ISRCTN13914201; EU-20613; EUDRACT-2005-001710-40
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer; Hypercalcemia of Malignancy; Metastatic Cancer
Keywords: hypercalcemia of malignancy; stage IV breast cancer; bone metastases; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Humoral Hypercalcemia Of Malignancy; Neoplasm Metastasis; Breast Neoplasms, Male | interventions — Ibandronic Acid; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibandronic Acid (Experimental): 50mg tablet once daily over 96 weeks
  Interventions: Drug: ibandronate sodium
- Zoledronic Acid (Active Comparator): 4 mg via intravenous infusion (iv) over a minimum of 15 minutes in at least 100mls of saline every 4 weeks over 96 weeks
  Interventions: Drug: zoledronic acid; Drug: Zolendronic Acid

INTERVENTIONS:
Drug: ibandronate sodium
  Arms: Ibandronic Acid
Drug: zoledronic acid
  Arms: Zoledronic Acid
Drug: Zolendronic Acid — Zoledronic acid 4 mg by intravenous infusion every 4 weeks.
  Other Names: Zoledronate
  Arms: Zoledronic Acid

SUMMARY:
RATIONALE: Ibandronate and zoledronate may help relieve some of the symptoms caused by bone metastases. It is not yet know whether ibandronate is more effective than zoledronate in treating bone metastases from breast cancer.

PURPOSE: This randomized phase III trial is studying ibandronate to see how well it works compared with zoledronate in treating patients with newly diagnosed bone metastases from breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy, in terms of reducing frequency and timing of skeletal-related events (SREs), of ibandronate vs zoledronate in patients with newly diagnosed bone metastases secondary to breast cancer.

Secondary

* Compare the median time to first SRE in patients treated with these regimens.
* Compare the percentage of patients experiencing a SRE after treatment with these regimens.
* Compare the number of occult vertebral fractures present in patients at the end of treatment with these regimens.
* Compare the pain and analgesic scores and quality of life of patients treated with these regimens.
* Compare the number of patients developing renal dysfunction or hypocalcemia during the study period.
* Compare the number of patients developing osteonecrosis of the jaw during study treatment and follow-up.
* Compare the overall survival of these patients at 96 weeks and at 5 years.
* Compare the health-resource usage of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, parallel-group, controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive zoledronate IV over 15 minutes on day 1. Treatment repeats every 21* or 28 days for at least 96 weeks (24 or 32 courses) in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients who receive concurrent chemotherapy every 3 weeks receive study treatment every 21 days

* Arm II: Patients receive oral ibandronate once daily on days 1-28. Treatment repeats every 28 days for at least 96 weeks (24 courses) in the absence of disease progression or unacceptable toxicity. Patients with bone pain or hypercalcemia at study entry or those who require IV therapy due to hypercalcemia while on study may receive 1 treatment with ibandronate IV at the discretion of the supervising clinician.

Quality of life and pain are assessed at baseline, after every 3 courses, and at completion of study treatment.

After completion of study treatment, patients are followed annually for up to 3 years.

PROJECTED ACCRUAL: A total of 1,400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven breast cancer

  * Metastatic disease
  * Previous relapsed disease in sites other than bone allowed
* Newly diagnosed multiple bone metastases within the past 3 months, meeting all of the following criteria:

  * Painful or asymptomatic
  * Lytic, mixed, or purely sclerotic type
  * Radiological diagnosis
  * IV bisphosphonate therapy indicated
* No CNS metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Male or female
* Menopausal status not specified
* No known active peptic ulcer
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active dental problems, including infection of the teeth or jawbone (maxilla or mandible) or dental or fixture trauma
* No prior or current diagnosis of osteonecrosis of the jaw, exposed bone in the mouth, or slow healing after dental procedures
* Creatinine clearance ≥ 30 mL/min
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* No history of bisphosphonate hypersensitivity
* Able to comply with instructions relating to oral study medications
* Able to take oral study medications
* No psychiatric illness or other condition that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* At least 6 months since prior bisphosphonate therapy
* At least 6 weeks since prior and no concurrent dental or jaw surgery (e.g., extractions or implants)

  * Concurrent unplanned dental extractions allowed provided study medication is discontinued for 8 weeks before and after the surgery
* Concurrent chemotherapy and/or hormone therapy for metastatic disease allowed
* No concurrent medications that affect bone metabolism (e.g., calcitonin or other nontrial bisphosphonates)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1404 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Frequency and timing of skeletal-related events (SREs) | 96 weeks

SECONDARY OUTCOMES:
Time to first SREs | 96 Weeks
Proportion of patients with SREs | 96 Weeks
Pain and analgesic score | 96 weeks
Quality of life | 96 weeks
Toxicity | 96 weeks
Survival | 5 years
Health resource usage and serum bone marker levels | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Barrett Lee, MD, Study Chair — Velindre NHS Trust
Locations (79):
- United Kingdom (79):
  - William Harvey Hospital, Ashford, England
  - North Devon District Hospital, Barnstaple, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Burnley General Hospital, Burnley, England
  - Queen's Hospital, Burton-on-Trent, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Countess of Chester Hospital, Chester, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Darent Valley Hospital, Dartford Kent, England
  - Derbyshire Royal Infirmary, Derby, England
  - Dorset County Hospital, Dorchester, England
  - University Hospital of North Durham, Durham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - Calderdale Royal Hospital, Halifax, England
  - University Hospital of Hartlepool, Hartlepool, Cleveland, England
  - Wycombe General Hospital, High Wycombe, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Ipswich Hospital, Ipswich, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Whipps Cross Hospital, London, England
  - Saint Bartholomew's Hospital, London, England
  - St. George's Hospital, London, England
  - Royal Marsden - London, London, England
  - Charing Cross Hospital, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - Maidstone Hospital, Maidstone, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Clatterbridge Centre for Oncology, Metropolitan Borough of Wirral, England
  - St. Mary's Hospital, Newport, England
  - Nottingham City Hospital, Nottingham, England
  - King's Mills Hospital, Nottinghamshire, England
  - George Eliot Hospital, Nuneaton, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Alexandra Healthcare NHS, Redditch, Worcestershire, England
  - Conquest Hospital, Saint Leonards-on-Sea, England
  - Scarborough General Hospital, Scarborough, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Solihull Hospital, Solihull, England
  - Southampton General Hospital, Southampton, England
  - University Hospital of North Tees, Stockton-on-Tees, England
  - Royal Marsden - Surrey, Sutton, England
  - Torbay Hospital, Torquay Devon, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - South Tyneside District Hospital, Tyne & Wear, England
  - Warrington Hospital NHS Trust, Warrington, England
  - South Warwickshire Hospital, Warwick, Warwickshire, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Royal Albert Edward Infirmary, Wigan, England
  - Royal Hampshire County Hospital, Winchester, England
  - Worcester Royal Hospital, Worcester, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Hairmyres Hospital, East Kilbride, Scotland
  - Falkirk and District Royal Infirmary, Falkirk, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Wishaw General Hospital, Wishaw, Scotland
  - Nevill Hall Hospital, Abergavenny, Wales
  - Bronglais District General Hospital, Aberystwyth, Wales
  - Ysbyty Gwynedd, Bangor, Wales
  - Princess of Wales Hospital, Bridgend, Wales
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - West Wales General Hospital, Carmarthen, Wales
  - Withybush General Hospital, Haverfordwest, Wales
  - Prince Charles Hospital, Mid Glamorgan, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - South West Wales Cancer Institute, Swansea, Wales
  - Wrexham Maelor Hospital, Wrexham, Wales
  - Royal Glamorgan Hospital, Llantrisant

REFERENCES:
- [Derived] Gillespie D, Farewell D, Barrett-Lee P, Casbard A, Hawthorne AB, Hurt C, Murray N, Probert C, Stenson R, Hood K. The use of randomisation-based efficacy estimators in non-inferiority trials. Trials. 2017 Mar 9;18(1):117. doi: 10.1186/s13063-017-1837-3. PMID 28274254
- [Derived] Barrett-Lee P, Casbard A, Abraham J, Hood K, Coleman R, Simmonds P, Timmins H, Wheatley D, Grieve R, Griffiths G, Murray N. Oral ibandronic acid versus intravenous zoledronic acid in treatment of bone metastases from breast cancer: a randomised, open label, non-inferiority phase 3 trial. Lancet Oncol. 2014 Jan;15(1):114-22. doi: 10.1016/S1470-2045(13)70539-4. Epub 2013 Dec 11. PMID 24332514